CLINICAL TRIAL: NCT02833844
Title: A Double Blind, Randomized, Placebo Controlled, Multicenter Study to Evaluate Safety, Tolerability, and Efficacy on LDL-C of Evolocumab (AMG 145) in Subjects With HIV and With Hyperlipidemia and/or Mixed Dyslipidemia
Brief Title: Safety, Tolerability and Efficacy on Low Density Lipoprotein Cholesterol (LDL-C) of Evolocumab in Participants With Human Immunodeficiency Virus (HIV) and Hyperlipidemia/Mixed Dyslipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20130286; 2015-004735-12 (EudraCT Number)
Record Dates: First submitted 2016-06-13; First posted 2016-07-14 (Estimated); Results first posted 2020-07-21 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Subjects With Hyperlipidemia, Dyslipidemia and HIV Infection
Keywords: Hyperlipidemia; Dyslipidemia; Proprotein convertase subtilisin/kexin type 9 (PCSK9); Inhibition; HIV infection; Cluster of differentiation; Viral load
MeSH Terms: conditions — Dyslipidemias; HIV Infections; Hyperlipidemias; Hypercholesterolemia, Autosomal Dominant, 3; Inhibition, Psychological | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Double-Blind Placebo SC QM/Open-Label Evolocumab 420 mg SC QM (Experimental): Double-blind placebo subcutaneous (SC) injection every 4 weeks (QM) for 24 weeks, followed by open-label evolocumab 420 mg SC QM for 24 weeks.
  Interventions: Drug: Evolocumab; Drug: Placebo
- Double-Blind Evolocumab 420 mg SC QM/Open-Label Evolocumab 420 mg SC QM (Placebo Comparator): Double-blind evolocumab SC injection QM for 24 weeks, followed by open-label evolocumab 420 mg SC QM for 24 weeks.
  Interventions: Drug: Evolocumab

INTERVENTIONS:
Drug: Evolocumab — Dose of subcutaneous evolocumab QM
  Other Names: EvoMab; Repatha; AMG 145
Drug: Placebo — Dose of matching placebo QM
  Arms: Double-Blind Placebo SC QM/Open-Label Evolocumab 420 mg SC QM

SUMMARY:
The study is divided into 2 parts. The first part of the study will be double-blinded and will last for 24 weeks. During this time, participants will be randomized in a ratio of 2:1 to receive either evolocumab once monthly (QM) or placebo QM. The second part of the study is a 24-week open label extension period. During this time all participants will receive evolocumab QM.

The clinical hypothesis is that subcutaneous evolocumab QM will be well tolerated and will result in greater reduction of low density lipoprotein cholesterol (LDL-C), defined as percent change from baseline at Week 24, compared with placebo QM in human immunodeficiency virus (HIV)-positive participants with hyperlipidemia or mixed dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Known HIV infection with stable HIV therapy for ≥ 6 months
* Cluster of differentiation 4 (CD4) ≥ 250 cells/mm^3 for ≥ 6 months
* HIV viral load ≤ 50 copies/mL at screening and ≤ 200 copies/mL for ≥ 6 months
* Subject on stable lipid-lowering therapy for ≥ 4 weeks prior to randomization and not expected to change during the duration of study
* For subjects with known clinical atherosclerotic cardiovascular disease (ASCVD), fasting LDL-C of ≥ 70 mg/dL or non-high density lipoprotein cholesterol (non-HDL-C) ≥ 100 mg/dL. For subjects without known clinical ASCVD: fasting LDL-C of ≥ 100 mg/dL or non-HDL-C of ≥ 130 mg/dL
* Fasting triglycerides ≤ 600 mg/dL (6.8 mmol/L)

Exclusion Criteria:

* Taking a combination of background lipid-lowering therapy and HIV therapy known to have significant drug-drug interaction
* New York Heart Association (NYHA) III or IV heart failure, or last known left ventricular ejection fraction (LVEF) < 30%
* Known opportunistic infection/acquired immunodeficiency syndrome (AIDS) defining illness within 1 year prior to randomization
* Myocardial infarction, unstable angina, percutaneous coronary intervention, coronary artery bypass graft or stroke within 3 months
* Type 1 diabetes, new-onset or poorly controlled type 2 diabetes
* Uncontrolled hypertension
* Taken a cholesteryl ester transfer protein inhibitor in the last 12 months
* Moderate to severe renal dysfunction
* Persistent active liver disease or hepatic dysfunction (Stable chronic hepatitis C of at least 1 year duration prior to randomization is allowed)
* Malignancy (except non-melanoma skin cancers, cervical in-situ carcinoma, breast ductal carcinoma in-situ, or stage 1 prostate carcinoma) within the last 5 years prior to randomization

Other exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2020-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (67):
- United States (18):
  - Research Site, Los Angeles, California
  - Research Site, Hartford, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Miami, Florida
  - Research Site, Tampa, Florida
  - Research Site, Vero Beach, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Berkley, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Southfield, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Camden, New Jersey
  - Research Site, Albany, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Falls Church, Virginia
- Australia (6):
  - Research Site, Darlinghurst, New South Wales
  - Research Site, East Sydney, New South Wales
  - Research Site, Sydney, New South Wales
  - Research Site, Fortitude Valley, Queensland
  - Research Site, Melbourne, Victoria
  - Research Site, Prahran, Victoria
- Belgium (3):
  - Research Site, Antwerp
  - Research Site, Brussels
  - Research Site, Ghent
- Brazil (3):
  - Research Site, São Paulo, São Paulo
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Canada (5):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- France (5):
  - Research Site, Bordeaux
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Paris
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- Italy (6):
  - Research Site, Bologna
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Pisa
  - Research Site, Roma
- Research Site, Warsaw, Poland
- Portugal (4):
  - Research Site, Almada
  - Research Site, Aveiro
  - Research Site, Coimbra
  - Research Site, Porto
- Romania (4):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Constanța
  - Research Site, Timișoara
- South Africa (3):
  - Research Site, Pretoria, Gauteng
  - Research Site, Westdene, Gauteng
  - Research Site, Bloemfontein
- Spain (2):
  - Research Site, Barcelona, Catalonia
  - Research Site, Madrid
- Switzerland (4):
  - Research Site, Geneva
  - Research Site, Lausanne
  - Research Site, Lugano
  - Research Site, Zurich
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Boccara F, Kumar PN, Caramelli B, Calmy A, Lopez JAG, Bray S, Cyrille M, Rosenson RS; BEIJERINCK Investigators. Evolocumab in HIV-Infected Patients With Dyslipidemia: Primary Results of the Randomized, Double-Blind BEIJERINCK Study. J Am Coll Cardiol. 2020 May 26;75(20):2570-2584. doi: 10.1016/j.jacc.2020.03.025. Epub 2020 Mar 28. PMID 32234462
- [Background] Boccara F, Kumar P, Caramelli B, Calmy A, Lopez JAG, Bray S, Cyrille M, Rosenson RS. Evolocumab treatment in patients with HIV and hypercholesterolemia/mixed dyslipidemia: BEIJERINCK study design and baseline characteristics. Am Heart J. 2020 Feb;220:203-212. doi: 10.1016/j.ahj.2019.11.004. Epub 2019 Nov 12. PMID 31841795
- [Background] Boccara F, Caramelli B, Calmy A, Kumar P, Lopez JAG, Bray S, Cyrille M, Rosenson RS; investigators of the BEIJERINCK study. Long-term effects of evolocumab in participants with HIV and dyslipidemia: results from the open-label extension period. AIDS. 2022 Apr 1;36(5):675-682. doi: 10.1097/QAD.0000000000003175. PMID 35025817
- [Derived] Schmidt AF, Carter JL, Pearce LS, Wilkins JT, Overington JP, Hingorani AD, Casas JP. PCSK9 monoclonal antibodies for the primary and secondary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2020 Oct 20;10(10):CD011748. doi: 10.1002/14651858.CD011748.pub3. PMID 33078867
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 72 centers in Australia, Belgium, Brazil, Canada, France, Greece, Italy, Poland, Portugal, Romania, South Africa, Spain, Switzerland, United Kingdom, and United States. The first participant was enrolled on 22 May 2017, and the last participant was enrolled on 23 January 2019.
Pre-assignment Details: Participants were randomized in a 2:1 ratio to evolocumab or placebo, respectively, in a double-blind manner. Randomization was stratified by entry statin treatment and hepatitis C status.
Groups:
- Double-Blind Placebo/Open-Label Evolocumab: Double-blind placebo subcutaneous (SC) injection every 4 weeks (QM) for 24 weeks in the double-blind period, followed by open-label evolocumab 420 mg SC QM for 24 weeks in the open-label period.
- Double-Blind Evolocumab/Open-Label Evolocumab: Double-blind evolocumab SC injection QM for 24 weeks in the double-blind period, followed by open-label evolocumab 420 mg SC QM for 24 weeks in the open-label period.
Period: Double-Blind Period
Arm/Group | Double-Blind Placebo/Open-Label Evolocumab | Double-Blind Evolocumab/Open-Label Evolocumab
Started (Randomized) | 157 | 310
Randomized and Treated | 157 | 307
Completed | 155 (completed double-blind period) | 303 (completed double-blind period)
Not Completed | 2 | 7
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Protocol Violation | 0 | 4
Period: Open-Label Period
Arm/Group | Double-Blind Placebo/Open-Label Evolocumab | Double-Blind Evolocumab/Open-Label Evolocumab
Started | 152 (3 participants did not continue to open-label period) | 303
Received Open-Label Study Drug | 152 | 299
Completed | 150 | 301
Not Completed | 2 | 2
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Double-Blind Placebo: Double-blind placebo SC injection QM for 24 weeks in the double-blind period.
- Double-Blind Evolocumab: Double-blind evolocumab SC injection QM for 24 weeks in the double-blind period.
- Total: Total of all reporting groups
Arm/Group | Double-Blind Placebo | Double-Blind Evolocumab | Total
Number analyzed (Participants) | 157 | 310 | 467
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (8.0) | 56.5 (9.1) | 56.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 45 | 82
  Male | 120 | 265 | 385
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 41 | 62
  Not Hispanic or Latino | 136 | 269 | 405
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 3 | 6
  Black or African American | 25 | 54 | 79
  White | 125 | 246 | 371
  Multiple Races | 1 | 0 | 1
  Other, Not Specified | 3 | 7 | 10
Stratification Factor: Statin Use at Baseline [Count of Participants; unit: Participants]
  Statin Use = Yes | 128 | 256 | 384
  Statin Use = No | 29 | 54 | 83
Stratification Factor: Hepatitis C Virus (HCV) Status at Baseline [Count of Participants; unit: Participants]
  HCV = Yes | 7 | 10 | 17
  HCV= No | 150 | 300 | 450
Low-Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] — Population: participants with a baseline assessment
  mg/dL
    number analyzed (Participants) | 157 | 306 | 463
    (all) | 133.26 (39.97) | 133.25 (40.25) | 133.25 (40.11)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in LDL-C at Week 24
Description: Least squares mean is from the repeated measures model which includes treatment group, statin stratification factor, scheduled visit and the interaction of treatment with scheduled visit as covariates. (Hepatitis C stratification factor is not included in the model due to low participant numbers.)
Time Frame: Baseline, Week 24
Population: Full Analysis Set: randomized participants who received at least 1 dose of investigational product. Participants with an assessment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- Double-Blind Placebo: Double-blind placebo SC injection QM for 24 weeks.
- Double-Blind Evolocumab: Double-blind evolocumab SC injection QM for 24 weeks.
Arm/Group | Double-Blind Placebo | Double-Blind Evolocumab
Number analyzed (Participants) | 151 | 295
percent change | 1.68 (2.03) | -55.23 (1.52)
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Evolocumab; Test type: Superiority; p < 0.0001, repeated measures linear effects model — Multiplicity adjustment was based on the combination of sequential testing, the fallback procedure, and the Hochberg procedure; Per protocol, the adjusted p-value is significant if less than the familywise error rate of 0.05; treatment difference = -56.92, 95% CI 2-sided [-61.55 to -52.28], Standard Error of Mean 2.36 — Treatment difference uses placebo as the reference

2. Secondary Outcome: Change From Baseline in LDL-C at Week 24
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Double-Blind Placebo | Double-Blind Evolocumab
Number analyzed (Participants) | 151 | 295
mg/dL | -2.3 (3.1) | -77.5 (2.3)
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Evolocumab; Test type: Superiority; p < 0.0001, repeated measures linear effects model — [p-value comment as in outcome 1, analysis 1]; Per protocol, the adjusted p-value is significant if less than the familywise error rate of 0.05; treatment difference = -75.2, 95% CI 2-sided [-82.1 to -68.4], Standard Error of Mean 3.5 — Treatment difference uses placebo as the reference

3. Secondary Outcome: Percentage of Participants Acheiving LDL-C < 70 mg/dL (1.8 mmol/L) at Week 24
Time Frame: Week 24
Population: Full Analysis Set: randomized participants who received at least 1 dose of investigational product. Participants with observed data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-Blind Placebo | Double-Blind Evolocumab
Number analyzed (Participants) | 151 | 296
percentage of participants | 7.9 [4.6 to 13.4] | 73.3 [68.0 to 78.0]
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Evolocumab; Multiplicity adjustment was based on the combination of sequential testing, the fallback procedure, and the Hochberg procedure; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Based on Cochran-Mantel-Haenszel test stratified by statin use stratification factor. For testing, nonachievement was imputed for participants with a missing value; Per protocol, the adjusted p-value is significant if less than the familywise error rate of 0.05; treatment difference = 65.4, 95% CI 2-sided [57.8 to 71.1] — Treatment difference uses placebo as reference

4. Secondary Outcome: Percentage of Participants With an LDL-C Response (50% Reduction of LDL-C From Baseline) at Week 24
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Double-Blind Placebo | Double-Blind Evolocumab
Number analyzed (Participants) | 151 | 295
percentage of participants | 0.7 [0.1 to 3.7] | 72.5 [67.2 to 77.3]
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Evolocumab; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Per protocol, the adjusted p-value is significant if less than the familywise error rate of 0.05; treatment difference = 71.9, 95% CI 2-sided [65.7 to 76.7] — Treatment difference uses placebo as a reference

5. Secondary Outcome: Percent Change From Baseline in Non-High-Density Lipoprotein Cholesterol (HDL-C) at Week 24
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Double-Blind Placebo | Double-Blind Evolocumab
Number analyzed (Participants) | 152 | 296
percent change | 2.86 (1.74) | -48.07 (1.31)
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Evolocumab; Test type: Superiority; p < 0.0001, repeated measures linear effects model — [p-value comment as in outcome 1, analysis 1]; Per protocol, the adjusted p-value is significant if less than the familywise error rate of 0.05; treatment difference = -50.94, 95% CI 2-sided [-54.88 to -46.99], Standard Error of Mean 2.01 — Treatment difference uses placebo as the reference

6. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (ApoB) at Week 24
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Double-Blind Placebo | Double-Blind Evolocumab
Number analyzed (Participants) | 153 | 302
percent change | 2.59 (1.50) | -45.14 (1.13)
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Evolocumab; Test type: Superiority; p < 0.0001, repeated measures linear effects model — [p-value comment as in outcome 1, analysis 1]; Per protocol, the adjusted p-value is significant if less than the familywise error rate of 0.05; treatment difference = -47.73, 95% CI 2-sided [-51.11 to -44.35], Standard Error of Mean 1.72 — Treatment difference uses placebo as the reference

7. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (TC) at Week 24
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Double-Blind Placebo | Double-Blind Evolocumab
Number analyzed (Participants) | 152 | 296
percent change | 2.34 (1.40) | -35.78 (1.06)
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Evolocumab; Test type: Superiority; p < 0.0001, repeated measures linear effects model — [p-value comment as in outcome 1, analysis 1]; Per protocol, the adjusted p-value is significant if less than the familywise error rate of 0.05; treatment difference = -38.12, 95% CI 2-sided [-41.30 to -34.94], Standard Error of Mean 1.62 — Treatment difference uses placebo as the reference

8. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) (Lp[a]) at Week 24
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Double-Blind Placebo | Double-Blind Evolocumab
Number analyzed (Participants) | 153 | 302
percent change | 10.35 (3.34) | -16.44 (2.57)
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Evolocumab; Test type: Superiority; p < 0.0001, repeated measures linear effects model — [p-value comment as in outcome 1, analysis 1]; Per protocol, the adjusted p-value is significant if less than the familywise error rate of 0.05; treatment difference = -26.78, 95% CI 2-sided [-34.17 to -19.40], Standard Error of Mean 3.76 — Treatment difference uses placebo as the reference

9. Secondary Outcome: Percent Change From Baseline in Triglycerides at Week 24
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Double-Blind Placebo | Double-Blind Evolocumab
Number analyzed (Participants) | 152 | 296
percent change | 13.21 (3.80) | -9.25 (2.89)
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Evolocumab; Test type: Superiority; p < 0.0001, repeated measures linear effects model — [p-value comment as in outcome 1, analysis 1]; Per protocol, the adjusted p-value is significant if less than the familywise error rate of 0.05; treatment difference = -22.46, 95% CI 2-sided [-31.03 to -13.88], Standard Error of Mean 4.36 — Treatment difference uses placebo as the reference

10. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 24
Description: as for outcome 1
Time Frame: Bseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Double-Blind Placebo | Double-Blind Evolocumab
Number analyzed (Participants) | 152 | 296
percent change | 2.73 (1.57) | 11.08 (1.20)
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Evolocumab; Test type: Superiority; p < 0.0001, repeated measures linear effects model — [p-value comment as in outcome 1, analysis 1]; Per protocol, the adjusted p-value is significant if less than the familywise error rate of 0.05; treatment difference = 8.36, 95% CI 2-sided [4.83 to 11.89], Standard Error of Mean 1.80 — Treatment difference uses placebo as the reference

11. Secondary Outcome: Percent Change From Baseline in Very Low-Density Lipoprotein Cholesterol (VLDL-C) at Week 24
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Double-Blind Placebo | Double-Blind Evolocumab
Number analyzed (Participants) | 141 | 284
percent change | 12.34 (3.54) | -9.81 (2.65)
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Evolocumab; Test type: Superiority; p < 0.0001, repeated measures linear effects model — [p-value comment as in outcome 1, analysis 1]; Per protocol, the adjusted p-value is significant if less than the familywise error rate of 0.05; treatment difference = -22.15, 95% CI 2-sided [-30.04 to -14.26], Standard Error of Mean 4.01 — Treatment difference uses placebo as the reference

ADVERSE EVENTS:
Time Frame: Double-blind Treatment (DBT) Period: From randomization (for all-cause mortality) or first dose of study drug (for adverse events) to up to week 24. Open-label Extension (OLE) Period: From the start of the OLE (week 24) to end of study (week 52) for all-cause mortality; and from first dose of study drug in the OLE up to 30 days after last dose, or end of study, whichever was earlier, for adverse events.
Description: Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug. All-cause mortality is reported for all participants randomized in the DBT Period as well as for all participants who entered into the OLE Period.
Groups:
- Double-Blind Placebo/Open-Label Evolocumab: Participants originally randomized to placebo in the double-blind period then received open-label evolocumab 420 mg SC QM for 24 weeks.
- Double-Blind Evolocumab/Open-Label Evolocumab: Participants originally randomized to evolocumab in the double-blind period then received open-label evolocumab 420 mg SC QM for 24 weeks.
Arm/Group | Double-Blind Placebo | Double-Blind Evolocumab | Double-Blind Placebo/Open-Label Evolocumab | Double-Blind Evolocumab/Open-Label Evolocumab
All-Cause Mortality (participants affected / at risk) | 0/157 | 0/310 | 0/152 | 2/303
Serious Adverse Events (participants affected / at risk) | 8/157 | 10/307 | 8/152 | 14/299
Other Adverse Events (participants affected / at risk) | 41/157 | 78/307 | 23/152 | 50/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Placebo (N=157) | Double-Blind Evolocumab (N=307) | Double-Blind Placebo/Open-Label Evolocumab (N=152) | Double-Blind Evolocumab/Open-Label Evolocumab (N=299)
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypertensive emergency (Vascular disorders) | 1 | 0 | 0 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1
Pericarditis constrictive (Cardiac disorders) | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Basosquamous carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hair follicle tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Renal cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Sarcomatoid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebral artery thrombosis (Nervous system disorders) | 0 | 0 | 1 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Placebo (N=157) | Double-Blind Evolocumab (N=307) | Double-Blind Placebo/Open-Label Evolocumab (N=152) | Double-Blind Evolocumab/Open-Label Evolocumab (N=299)
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 11 | 1 | 8
Chest pain (General disorders) | 5 | 2 | 0 | 1
Influenza like illness (General disorders) | 4 | 12 | 2 | 3
Nasopharyngitis (Infections and infestations) | 2 | 10 | 6 | 9
Upper respiratory tract infection (Infections and infestations) | 4 | 7 | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 9 | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 12 | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 6 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 7 | 0 | 1
Headache (Nervous system disorders) | 5 | 6 | 3 | 1
Paraesthesia (Nervous system disorders) | 0 | 7 | 0 | 1
Hypertension (Vascular disorders) | 5 | 0 | 3 | 4
Bronchitis (Infections and infestations) | 3 | 5 | 2 | 7
Sinusitis (Infections and infestations) | 1 | 1 | 1 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT02833844/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT02833844/SAP_001.pdf